CLINICAL TRIAL: NCT01433536
Title: Evaluation of Circulating Osteogenic Factors in Trauma Patients (BMP-9)
Brief Title: Evaluation of Circulating Osteogenic Factors in Trauma Patients
Acronym: BMP-9
Status: Terminated | Type: Observational
Why Stopped: Guillaume Grenier, principal investigator is no longer working at the lab. The lab is now closed.
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Collaborators: Université de Sherbrooke (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Guillaume Grenier, Associate Professor, Université de Sherbrooke
Other Study IDs: 10-100; MOP-115149 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2011-09-12; First posted 2011-09-14 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Healthy; High Velocity Fracture; Cranial Trauma; Spinal Trauma
Keywords: cranial trauma with or without high velocity fracture to inferior limb; spinal trauma with or without high velocity fracture to inferior limb; high velocity fracture to inferior limb

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- cranial trauma and fracture: Individuals presenting a cranial trauma that are classified at equal to or less than 8 on the Glasgow scale, combined with a fracture to the femur, tibia, or pelvis resulting from a high-velocity impact
- cranial trauma: Individuals presenting a cranial trauma that are classified at equal to or less than 8 on the Glasgow scale
- spinal trauma with fracture: Individuals presenting a spinal fracture that are classified with an ASIA score of A, B, or C, combined with a fracture to the femur, tibia, or pelvis resulting from a high-velocity impact
- spinal trauma: Individuals presenting a spinal fracture that are classified with an ASIA score of A, B, or C
- high velocity fracture, inferior limb: Individuals that present a fracture to the femur, tibia, or pelvis resulting from a high-velocity impact
- Control: Healthy individuals

SUMMARY:
Bone fractures in traumatic brain-injured and spinal cord-injured patients often heal faster than in other patients. However, such patients are also occasionally prone to bone formation in soft tissues such as muscle. This process is called heterotopic ossification and tends to occur around joints. Patients with heterotopic ossification often suffer from complications such nerve compression, ankylosis, chronic pain, osteoporosis, and infections. Loss of movement can also interfere with function and the quality of life of patients already experiencing difficulties associated with their trauma. Positioning, transfers, and hygiene become difficult and even impossible, which worsens the loss of autonomy.

Previous research has suggested that an osteoinductive factor (which has the capacity to induce the formation of bone) may be released into the bloodstream following a head or spinal cord injury. The investigators laboratory has shown that a growth factor called BMP-9, when injected into a damaged mouse muscle, has the ability to cause strong ossification in damaged muscle. The investigators would like to find out whether the levels of BMP-9 and/or its receptor (which is called ALK1) increase after traumatic brain and spinal cord injuries that occur at the same time as serious orthopaedic traumas.

The main goal of the investigators study is thus to determine whether BMP-9 levels increase in the serum of trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* cranial trauma with Glasgow =< 8
* spinal trauma with ASIA A, B, C
* high-velocity fracture of femur, tibia, pelvis

Exclusion Criteria:

* brain dead
* pathological fractures (cancer, osteoporosis)
* blood transfusion received
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients arriving at the emergency room at the CHUS that present pathologies associated with the different cohorts described and responding to inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-12; Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Grenier, Ph.D., Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided